CLINICAL TRIAL: NCT02215668
Title: Impact of Physical Exercise, Aimed at Reducing Pain in Women Who Underwent Mammography.
Brief Title: The Effect of Physical Exercise in Reducing Pain in Women Undergoing Mammography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Altacílio Aparecido Nunes, Full professor; MD; Ph.D., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 313.907
Record Dates: First submitted 2014-08-09; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Pain; Side Effects
MeSH Terms: conditions — Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No physical exercise (No Intervention): Women are never subjected to any exercise prior to mammography.
- Physical exercise (Upper limb) (Experimental): Women will be subjected to physical exercise on upper limb prior to mammography.
  Interventions: Procedure: Physical exercise
- Group 2 (Active Comparator): Women are subjected to physical exercise in the lower limbs prior to mammography
  Interventions: Procedure: Physical exercise

INTERVENTIONS:
Procedure: Physical exercise — Exercise muscle stretching and body warming.
  Other Names: Physical activity
  Arms: Group 2; Physical exercise (Upper limb)

SUMMARY:
Mammography is a systematic way in the main programs of screening for breast cancer in women over 40 or 50 years old, according to screening programs, but most research has shown a frequency of discomfort and pain during the examination mammography. This study is a randomized controlled trial, whose intervention will be a sequence of exercises body warming and muscle stretching, performed systematic manner and supervised by a physical educator. It is expected to find in this study a possible impact of physical exercise in reducing pain after mammography examination.

DETAILED DESCRIPTION:
This research aims to evaluate the relationship of pre-mammography guided physical activity and pain after the examination, evaluating the impact of the intervention in a group of patients undergoing upper limb exercise (SLE), compared to another group women not subject exposure (MNE), and another group with lower limb exercise (LLE). This study is a randomized controlled trial, whose intervention will be a sequence of exercises body warming and muscle stretching, performed systematic manner and supervised by a physical educator. It is expected to find in this study a possible impact of physical exercise in reducing pain after mammography examination. The results will be checked by study association between the level of physical activity, body mass index, breast density and reducing the pain effect between groups for comparison of means and variances of values of the visual analogue scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Women: 20 to 69 years old

Exclusion Criteria:

* Cardiovascular disease
* Mental diseases
* Pulmonary diseases
* Steroids use

Ages: 20 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Decreased pain after mammography. | Decrease in pain after performing mammography, checked10 minutes after the procedure e, measured by visual analog scale.
  Following the randomization, approximately 10 minutes after performing a physical exercise in the upper limbs (Group 1) and lower (Group 2), or not performing any physical exercise (Group 0), the woman will be submitted to bilateral mammogram. Ten minutes after the procedure, the assessment of pain during mammography will be measured by the visual analog scale. The mean difference between the measurements of visual analog scale (VAS) will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Altacilio A Nunes, MD; Ph.D, Principal Investigator — Ribeirao Preto Medical School - USP
Locations (1):
- Hospital do Cancer de Barretos, Barretos, São Paulo, Brazil